CLINICAL TRIAL: NCT05606809
Title: Comparison of Scores for Early Brain Damage Assessment at Intensive Care Unit Admission After Cardiac Arrest
Acronym: AfterROSC2
Status: Recruiting | Type: Observational
Sponsor: AfterROSC (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01811-42
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; intensive care unit; mechanical ventilation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Calculation of early prognosis score — Early prognosis score will be calculated at intensive care unit admission for each patient based on clinical and biological values as required

SUMMARY:
Even in patients with successful return of spontaneous circulation (ROSC), outcome after cardiac arrest remains poor. The overall in-hospital survival rate widely varies both worldwide and across communities, from 1 to 4 folds according to circumstances of arrest and post-resuscitation interventions. Several studies have already shown that early interventions performed after ROSC, such as treatment of the cause, targeted temperature management, optimal hemodynamic management and extra-corporeal life support in selected patients, could improve the outcome in post-cardiac arrest patients. However, the decision process regarding the allocation of these resources, in parallel with the management of patients' proxies, remains a complex challenge for physicians facing these situations. Consequently, several prediction models and scores have been developed in order to stratify the risk of unfavorable outcome and to discriminate the best candidates for post-resuscitation interventions. Overall, several scores exist, but external validation are lacking and direct comparisons are needed to assess relative interest of scoring systems. Indeed, establishing the optimal scoring system is crucial, for optimal treatment allocation and appropriate information to relatives.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients, major, admitted to intensive care after cardiac arrest (after both in and out-of hospital cardiac arrest),
* comatose (defined by Glasgow score ≤ 8) on admission,

Exclusion Criteria:

* cardiac arrest occurring intra-hospital,
* minor patient,
* major patient under guardianship,
* protected persons,
* prior inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational, prospective, multicentric prognostic study. The study period is 3 years, and investigators plan to include 4500 patients in 20 ICUs in France.
  For all patients included, medical history, clinical data, paraclinical results and outcome (at hospital discharge and at 3 months, including modified Rankin score) will be prospectively collected by local investigator, according to an electronical CRF.
Sampling Method: Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Determination of Area Under Curve of Cerebral Admission Hospital Prognosis (CAHP) Score at intensive care unit admission | Intensive Care Unit Admission (Usually 3 hours after cardiac arrest
  Determination of AUC for CAHP score as compare to Utstein style criteria.
  CAHP score range from 0 to 300 with higher score indicates poorer prognosis

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU Nantes, Nantes, Pays de Loire
  - Hopital Jacques Cartier, Massy
  - Clinique Ambroise Paré, Neuilly-sur-Seine
  - APHP, Cochin, Paris
  - CH Versailles, Versailles

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of IPD will be possible upon request to steering committee of the AfterROSC Network after approval of the project by ethics committee.